CLINICAL TRIAL: NCT00002434
Title: A Study of Trimetrexate Glucuronate (Neutrexin) With Leucovorin Protection for Patients With Pneumocystis Carinii Pneumonia
Brief Title: A Study of Neutrexin Plus Leucovorin in the Treatment of Pneumocystis Carinii Pneumonia (PCP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: U.S. Bioscience (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 132A; TMTX 0014
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1994-01

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Trimetrexate; Pneumonia, Pneumocystis carinii; Leucovorin; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — trimetrexate glucuronate; Leucovorin

INTERVENTIONS:
Drug: Trimetrexate glucuronate
Drug: Leucovorin calcium

SUMMARY:
To evaluate the safety and efficacy of trimetrexate glucuronate with leucovorin protection in patients with Pneumocystis carinii pneumonia (PCP) who are refractory to or have demonstrated severe or life-threatening toxicities to standard therapies (e.g., TMP/SMX or parenteral pentamidine).

DETAILED DESCRIPTION:
Patients receive intravenous infusions of trimetrexate glucuronate and leucovorin for 21 days. Leucovorin is continued for 3 additional days after discontinuation of trimetrexate glucuronate. Patients are followed for 1 month.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Myelosuppressive or nephrotoxic agents at the discretion of the treating physician.

Patients must have:

* Pneumocystis carinii pneumonia (PCP) confirmed within 15 days prior to study entry.
* Serious intolerance and/or resistance to standard therapies (such as trimethoprim/sulfamethoxazole and parenteral pentamidine) during the course of therapy for the current episode of PCP, or a documented history of such intolerance during a prior episode.
* Consent of parent or guardian if less than 18 years of age.

NOTE:

* Pregnant women may enroll after the physician and patient have discussed the potential benefit versus risk.

Exclusion Criteria

Patients with the following prior conditions are excluded:

History of Type I hypersensitivity (i.e., urticaria, angioedema, or anaphylaxis), exfoliative dermatitis, or other life-threatening reactions due to trimetrexate glucuronate.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Feinberg J, Study Chair
Locations (1):
- United States Bioscience Inc, West Conshohocken, Pennsylvania, United States

REFERENCES:
- [Background] Feinberg J, McDermott C, Nutter J. Trimetrexate (TMTX) salvage therapy for PCP in AIDS patients with limited therapeutic options. Int Conf AIDS. 1992 Jul 19-24;8(2):B136 (abstract no PoB 3297)